## Informed Consent Form:

## "Treatment of impending ulcers associated with hammer, mallet and claw toe deformities in the diabetic patient setting"

## **Declaration from research participant:**

I have received sufficient written and oral information regarding aim, method, advantages and risks to agree to participation in this project

I am conscious that participation is voluntary, and that I can always retract my consent, without giving up my current or future rights in relation to treatment.

I hereby consent to participation in this research project and have been offered a copy of the consent form and the written information regarding this project.

| Research participants name: | |
|---|---|
| Patient ID Number | er: |
| Date: | Signature: |
| | related information regarding, you is discovered during the course of the project you If you do <b>not</b> wish to be informed, please mark with x here: |
| Do you wish to b to your treatmen | e informed on results of the project after conclusion of the project, and how it pertains t: |
| Yes | No |
| Declaration fro | m investigator who supplied information: |
| I hereby declare | that participant has received written and oral information pertaining to the project. |
| To the best of my participation in the | y knowledge the given information is sufficient for participant to make decision regarding<br>ne project. |
| Name of the inve | stigator that has given the information: |
| Date: | Signature: |

Version 1.2 Page 1